CLINICAL TRIAL: NCT04382404
Title: Phase 1 Pharmacokinetic Trial of Sofosbuvir/Velpatasvir in Pregnant Women With Chronic Hepatitis C Virus Infection
Brief Title: Treatment of Chronic Hepatitis C During Pregnancy With Sofosbuvir/Velpatasvir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Anne Chappell (Other)
Collaborators: Gilead Sciences (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Catherine Anne Chappell, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100377; R21HD101996 (NIH)
Record Dates: First submitted 2020-02-16; First posted 2020-05-11 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis C, Chronic
Keywords: pregnancy
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Intervention Model Description: Open-label, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sofosbuvir-Velpatasvir (Experimental): Sofosbuvir-Velpatasvir
  Interventions: Drug: Sofosbuvir-Velpatasvir Drug Combination

INTERVENTIONS:
Drug: Sofosbuvir-Velpatasvir Drug Combination — One oral pill containing 400mg sofosbuvir and 100mg velpatasvir taken once daily for 12 weeks
  Other Names: Epclusa

SUMMARY:
A single-arm, single-center, open label Phase 1 study of a 12-week course of Sofosbuvir (SOF)/Velpatasvir (VEL) in 10 HCV-infected pregnant women 1 that will evaluate the plasma pharmacokinetic parameters of SOF/VEL administered during pregnancy and compare them to those of a historical cohort of nonpregnant women.

DETAILED DESCRIPTION:
A single-arm, single-center, open label Phase 1 study of a 12-week course of SOF/VEL in 10 HCV-infected pregnant women. Treatment will be initiated during the second trimester, reducing the risk of SOF/VEL exposure during organogenesis and ensuring treatment completion by delivery, minimizing the risk of perinatal transmission. The study will be completed in 10 or 11 visits (7 maternal visits, delivery visit and 3 infant visits) which should align with prenatal and postpartum visits. Patients will be screened between 14+0 and 22+6 weeks of gestation confirmed by ultrasound by the time of their enrollment visit who are known to have chronic HCV infection. An HCV RNA level to confirm the patient is actively infected with HCV as well as an HCV genotype will be obtained. A full laboratory evaluation of liver function will be obtained to evaluate for renal failure and decompensated cirrhosis. A Hepatitis B Virus (HBV) panel will be performed to test all patients for evidence of current or prior HBV infection before initiation of HCV treatment. If the inclusion and exclusion criteria are met, the patient will be enrolled into the study between 23+0 and 25+6 weeks' gestation and initiated on a 12 week course of SOF/VEL. Systemic exposure of both VEL and SOF (SOF and inactive metabolite GS-331007) and intracellular SOF (GS-461203) will be assessed by pharmacokinetic sampling at 3, 6, and 9 weeks after first dose. HCV RNA viral load will be assessed at 12 weeks after completion of SOF/VEL treatment. Pregnancy and delivery outcomes will be collected prospectively. Neonatal outcomes will be assessed at birth, 8 weeks, 6 months and 12 months. HCV RNA viral load will be obtained at birth (as available), 1 to 3 months, at 6 months and then again at 12 months only if negative viral loads are not documented at 1 to 3 and 6 months. Neurodevelopmental assessments will be obtained at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and take part in the study -procedures
* Able and willing to provide adequate locator information
* Chronic hepatitis C viral (HCV) infection, defined as a positive HCV test at least 6 months prior to screening
* Detectable HCV RNA viral load at Screening
* Desired pregnancy at 23 + 0 to 25 + 6 weeks' gestation at enrollment with gestational dating confirmed by ultrasound
* Singleton gestation with no known fetal abnormalities
* Documented negative Hepatitis B (HB) testing for current infection (negative HB serum antigen test) or previous infection (negative anti-HB Core) performed at the screening visit
* Negative HIV testing at the screening visit
* Per participant report at screening and enrollment, agrees not to participate in other research studies involving drugs or medical devices for the duration of study participation

Exclusion Criteria:

* Participant report of any of the following at screening or enrollment:

  1. Previous treatment for Hepatitis C virus with sofosbuvir or a non-structural protein 5A inhibitor
  2. Use of any medications contraindicated with concurrent use of velpatasvir or sofosbuvir according to the most current Epclusa package insert
  3. Plans to relocate away from the study site area in the next 1 year and 4 months and unable/unwilling to return for study visits
  4. Current sexual partner is known to be infected with HIV or Hepatitis B virus
  5. History of cirrhosis documented or reported by previous liver biopsy or liver imaging tests
* Reports participating in any other research study involving drugs or medical devices within 60 days or less prior to enrollment
* Clinically significant and habitual non-therapeutic drug abuse, not including marijuana, as determined by Protocol Chair
* At Screening or Enrollment, as determined by the Protocol Chair, any significant uncontrolled active or chronic cardiovascular, renal, liver (such as evidence of decompensated cirrhosis by ascites, encephalopathy, or variceal hemorrhage), hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease (other than Hepatitis C)
* Has a high risk of preterm birth defined as a history of spontaneous preterm birth at less than 34 weeks of gestation or a shortened cervical length of less than 20 millimeters
* Has any of the following laboratory abnormalities at screening:

  1. Aspartate aminotransferase or alanine transaminase greater than 10 times the upper limited of normal
  2. Hemoglobin less than 9g/dL
  3. Platelet count less than 90,000 per mm3
  4. International normalized ratio > 1.5
  5. Creatinine greater than 1.4
* Has any other condition that, in the opinion of the investigator or designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chappell, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be submitted by email to the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after the primary manuscript for the study is published. Information will be available for an indefinite period of time.
Access Criteria: Data requests submitted by email will be reviewed by the Principal Investigator on a case by case basis.

REFERENCES:
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Hughes BL, Page CM, Kuller JA. Hepatitis C in pregnancy: screening, treatment, and management. Am J Obstet Gynecol. 2017 Nov;217(5):B2-B12. doi: 10.1016/j.ajog.2017.07.039. Epub 2017 Aug 4. PMID 28782502
- [Background] Gilbert EM, Darin KM, Scarsi KK, McLaughlin MM. Antiretroviral Pharmacokinetics in Pregnant Women. Pharmacotherapy. 2015 Sep;35(9):838-55. doi: 10.1002/phar.1626. Epub 2015 Aug 21. PMID 26297552
- [Background] Chappell CA, Krans EE, Bunge KE, Macio IS, Bogen D, Scarsi KK, Meyn LA, Hillier SL. A Phase 1 Study of Ledipasvir/Sofosbuvir in Pregnant Women with Hepatitis C Virus. In: Conferences on Retroviruses and Opportunistic Infections; 2010 Mar 4-7; Seattle, WA; Abstract 87
- [Background] Ward RM, Varner MW. Principles of Pharmacokinetics in the Pregnant Woman and Fetus. Clin Perinatol. 2019 Jun;46(2):383-398. doi: 10.1016/j.clp.2019.02.014. Epub 2019 Mar 30. PMID 31010566
- [Background] MacBrayne CE, Kiser JJ. Pharmacologic Considerations in the Treatment of Hepatitis C Virus in Persons With HIV. Clin Infect Dis. 2016 Jul 15;63 Suppl 1(Suppl 1):S12-23. doi: 10.1093/cid/ciw220. PMID 27363437
- [Background] Kirby BJ, Symonds WT, Kearney BP, Mathias AA. Pharmacokinetic, Pharmacodynamic, and Drug-Interaction Profile of the Hepatitis C Virus NS5B Polymerase Inhibitor Sofosbuvir. Clin Pharmacokinet. 2015 Jul;54(7):677-90. doi: 10.1007/s40262-015-0261-7. PMID 25822283
- [Background] Feld JJ, Jacobson IM, Hezode C, Asselah T, Ruane PJ, Gruener N, Abergel A, Mangia A, Lai CL, Chan HL, Mazzotta F, Moreno C, Yoshida E, Shafran SD, Towner WJ, Tran TT, McNally J, Osinusi A, Svarovskaia E, Zhu Y, Brainard DM, McHutchison JG, Agarwal K, Zeuzem S; ASTRAL-1 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 1, 2, 4, 5, and 6 Infection. N Engl J Med. 2015 Dec 31;373(27):2599-607. doi: 10.1056/NEJMoa1512610. Epub 2015 Nov 16. PMID 26571066
- [Background] Foster GR, Afdhal N, Roberts SK, Brau N, Gane EJ, Pianko S, Lawitz E, Thompson A, Shiffman ML, Cooper C, Towner WJ, Conway B, Ruane P, Bourliere M, Asselah T, Berg T, Zeuzem S, Rosenberg W, Agarwal K, Stedman CA, Mo H, Dvory-Sobol H, Han L, Wang J, McNally J, Osinusi A, Brainard DM, McHutchison JG, Mazzotta F, Tran TT, Gordon SC, Patel K, Reau N, Mangia A, Sulkowski M; ASTRAL-2 Investigators; ASTRAL-3 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 2 and 3 Infection. N Engl J Med. 2015 Dec 31;373(27):2608-17. doi: 10.1056/NEJMoa1512612. Epub 2015 Nov 17. PMID 26575258
- See also: Food and Drug Administration. Epclusa Package Insert. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2016/208341s000lbl.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 mother-infant dyads were enrolled
Groups:
- Sofosbuvir-Velpatasvir: One oral pill containing 400mg sofosbuvir and 100mg velpatasvir taken once daily for 12 weeks
Period: Overall Study
Arm/Group | Sofosbuvir-Velpatasvir
Started | 11 (Mothers: 11 participants; Infants: 11 participants)
Completed | 8 (Mothers: 8 participants; Infants: 8 participants)
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Maternal baseline characteristics are reported unless otherwise stated
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] — Population: Age in years reported for 11 maternal participants
  years
    Maternal Age, years: number analyzed (Participants) | 11
    Maternal Age, years | 30 [25 to 39]
Age, Continuous [Median (Full Range); unit: weeks] — Population: Age in weeks reflects gestational age of the 11 infant participants at birth
  weeks
    Infant Age, weeks: number analyzed (Participants) | 11
    Infant Age, weeks | 39.00 [35.57 to 39.43]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex of maternal and infant participants reported separately
  Participants
    Mothers: number analyzed (Participants) | 11
    Mothers: Female | 11
    Mothers: Male | 0
    Infants: number analyzed (Participants) | 11
    Infants: Female | 6
    Infants: Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity of maternal and infant participants reported separately
  Participants
    Mothers: number analyzed (Participants) | 11
    Mothers: Hispanic or Latino | 0
    Mothers: Not Hispanic or Latino | 11
    Mothers: Unknown or Not Reported | 0
    Infants: number analyzed (Participants) | 11
    Infants: Hispanic or Latino | 1
    Infants: Not Hispanic or Latino | 10
    Infants: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race of maternal and infant participants reported separately
  Participants
    Mothers: number analyzed (Participants) | 11
    Mothers: American Indian or Alaska Native | 0
    Mothers: Asian | 0
    Mothers: Native Hawaiian or Other Pacific Islander | 0
    Mothers: Black or African American | 1
    Mothers: White | 10
    Mothers: More than one race | 0
    Mothers: Unknown or Not Reported | 0
    Infants: number analyzed (Participants) | 11
    Infants: American Indian or Alaska Native | 0
    Infants: Asian | 0
    Infants: Native Hawaiian or Other Pacific Islander | 0
    Infants: Black or African American | 1
    Infants: White | 9
    Infants: More than one race | 1
    Infants: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Hepatitis C Virus Genotype [Count of Participants; unit: Participants] — Population: Data only relevant to maternal participants
  Participants
    number analyzed (Participants) | 11
    Genotype 1 | 8
    Genotype 3 | 3
Gestational Age at Treatment Start [Median (Full Range); unit: weeks] — Population: Data only relevant to maternal participants
  weeks
    number analyzed (Participants) | 11
    (all) | 23.43 [23.00 to 25.86]
Weight [Median (Full Range); unit: kg] — Population: Weight reported separately for maternal and infant participants
  kg
    Mothers: number analyzed (Participants) | 11
    Mothers | 73.5 [54.4 to 101.1]
    Infants: number analyzed (Participants) | 11
    Infants | 2.9 [2.5 to 3.8]
Body Mass Index [Median (Full Range); unit: kg/m2] — Population: Body mass index only measured for maternal participants
  kg/m2
    number analyzed (Participants) | 11
    (all) | 27.0 [22.7 to 34.9]
Serum Creatinine [Median (Full Range); unit: mg/dL] — Population: Data only measured in maternal participants
  mg/dL
    number analyzed (Participants) | 11
    (all) | 0.5 [0.4 to 0.6]
Hematocrit [Median (Full Range); unit: percent] — Population: Data only measured in maternal participants
  percent
    number analyzed (Participants) | 11
    (all) | 36 [33 to 38]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration of Velpatasvir in Maternal Plasma
Description: Maximum concentration of Velpatasvir measured in maternal plasma samples. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation. At the 6-week visit, a single convenience blood sample was collected.
Time Frame: Up to 9 weeks from initiation of treatment
Population: 10 maternal participants had results from 2 or more visits; 1 maternal participant discontinued study drug after one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
ng/mL | 381.93 (38.35)
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; Maximum concentration of Velpatasvir in plasma was compared between the 10 pregnant women in this study to 25 non-pregnant historical control women. The geometric mean concentration (percent coefficient of variation) for the non-pregnant cohort was 449.39 (77.12); Test type: Other; Geometric mean ratio = 0.85, 90% CI 2-sided [0.63 to 1.15] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

2. Primary Outcome: Maximum Concentration of Sofosbuvir in Maternal Plasma
Description: Maximum concentration of Sofosbuvir measured in maternal plasma samples. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation. At the 6-week visit, a single convenience blood sample was collected.
Time Frame: Up to 9-weeks from initiation of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
ng/mL | 1455.09 (43.92)
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; Maximum concentration of Sofosbuvir in plasma was compared between the 10 pregnant women in this study to 25 non-pregnant historical control women. The geometric mean concentration (percent coefficient of variation) for the non-pregnant cohort was 1226.16 (59.46); Test type: Other; Geometric mean ratio = 1.19, 90% CI 2-sided [0.88 to 1.60] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

3. Primary Outcome: Maximum Concentration of GS-331007 in Maternal Plasma
Description: Maximum concentration of GS-331007, an inactive metabolite of Sofosbuvir, measured in maternal plasma samples. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation. At the 6-week visit, a single convenience blood sample was collected.
Time Frame: Up to 9 weeks from initiation of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
ng/mL | 752.66 (21.85)
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; Maximum concentration of GS-331007 in plasma was compared between the 10 pregnant women in this study to 25 non-pregnant historical control women. The geometric mean concentration (percent coefficient of variation) for the non-pregnant cohort was 1312.17 (32.55); Test type: Other; Geometric mean ratio = 0.57, 90% CI 2-sided [0.49 to 0.67] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

4. Primary Outcome: Area Under the Maternal Plasma Concentration Versus Time Curve of Velpatasvir
Description: Area under the maternal plasma concentration of Velpatasvir versus time curve tau of the dosing interval. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation.
Time Frame: Up to 9 weeks from initiation of treatment
Population: 10 participants had results from 2 or more visits; 1 participant discontinued study drug after one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
hr*ng/mL | 3244.45 (39.89)
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; Area under the plasma concentration versus time curve tau of Velpatasvir was compared between the 10 pregnant women in this study to 25 non-pregnant historical control women. The geometric mean (percent coefficient of variation) for the non-pregnant cohort was 3570.65 (72.04); Test type: Other; Geometric mean ratio = 0.91, 90% CI 2-sided [0.67 to 1.23] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

5. Primary Outcome: Area Under the Maternal Plasma Concentration Versus Time Curve of Sofosbuvir
Description: Area under the maternal plasma concentration of Sofosbuvir versus time curve tau of the dosing interval. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation.
Time Frame: Up to 9 weeks from initiation of treatment
Population: 10 participants had results from 2 or more visits; 1 participant discontinued study drug after one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
hr*ng/mL | 2039.62 (29.75)
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; Area under the plasma concentration versus time curve tau of Sofosbuvir was compared between the 10 pregnant women in this study to 25 non-pregnant historical control women. The geometric mean (percent coefficient of variation) for the non-pregnant cohort was 1483.83 (66.43); Test type: Other; Geometric mean ratio = 1.39, 90% CI 2-sided [1.06 to 1.78]; The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

6. Primary Outcome: Area Under the Maternal Plasma Concentration Versus Time Curve of GS-331007
Description: Area under the maternal plasma concentration of GS-331007 versus time curve tau of the dosing interval; GS-331007 is an inactive metabolite of Sofosbuvir. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation.
Time Frame: Up to 9 weeks from initiation of treatment
Population: 10 participants had results from 2 or more visits; 1 participant discontinued study drug after one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
hr*ng/mL | 9558.94 (18.75)
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; Area under the plasma concentration versus time curve tau of Sofosbuvir was compared between the 10 pregnant women in this study to 25 non-pregnant historical control women. The geometric mean (percent coefficient of variation) for the non-pregnant cohort was 15361.31 (22.35); Test type: Other; Geometric mean ratio = 0.62, 90% CI 2-sided [0.55 to 0.71]; The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

7. Secondary Outcome: Intracellular Concentration of GS-461203 From Maternal Peripheral Blood Mononuclear Cells at 3 Weeks
Description: Intracellular concentration of GS-461203, the active form of Sofosbuvir, from maternal peripheral blood mononuclear cells measured 3 weeks after initiation of treatment
Time Frame: Approximately 3 weeks from initiation of treatment
Population: One participant discontinued study medication after the second daily dose
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/10^6 cells
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
fmol/10^6 cells | 2111 [1096 to 4066]
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; The geometric mean (95 percent confidence interval) concentration of GS-461203 in peripheral blood mononuclear cells was compared between the pregnant cohort and 58 nonpregnant persons. The geometric mean (95 percent confidence interval) concentration of GS-461203 was 1474 (488, 4453) fmol /10^6 cells in the nonpregnant cohort; Test type: Other; Geometric mean ratio = 1.43, 95% CI 2-sided [0.91 to 2.25]; The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

8. Secondary Outcome: Intracellular Concentration of GS-461203 From Maternal Peripheral Blood Mononuclear Cells at 6 Weeks
Description: Intracellular concentration of GS-461203, the active form of Sofosbuvir, from maternal peripheral blood mononuclear cells measured 6 weeks after initiation of treatment
Time Frame: Approximately 6 weeks from initiation of treatment
Population: One participant discontinued study medication after the second daily dose
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/10^6 cells
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
fmol/10^6 cells | 2808 [1559 to 5058]
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; [analysis description as in outcome 7, analysis 1]; Test type: Other; Geometric mean ratio = 1.91, 95% CI 2-sided [1.14 to 3.19] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

9. Secondary Outcome: Intracellular Concentration of GS-461203 From Maternal Peripheral Blood Mononuclear Cells at 9 Weeks
Description: Intracellular concentration of GS-461203, the active form of Sofosbuvir, from maternal peripheral blood mononuclear cells measured 9 weeks after initiation of treatment
Time Frame: Approximately 9 weeks from initiation of treatment
Population: One participant discontinued study medication after the second daily dose
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/10^6 cells
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
fmol/10^6 cells | 2212 [1267 to 3864]
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; [analysis description as in outcome 7, analysis 1]; Test type: Other; Geometric mean ratio = 1.50, 95% CI 2-sided [0.87 to 2.60] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

10. Secondary Outcome: Intracellular Concentration of GS-461203 From Dried Maternal Blood Spots at 3 Weeks
Description: Intracellular concentration of GS-461203, the active form of Sofosbuvir, from dried maternal blood spots measured 3 weeks after initiation of treatment
Time Frame: Approximately 3 weeks from initiation of treatment
Population: One participant discontinued study medication after the second daily dose
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/punch
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
fmol/punch | 340 [287 to 403]
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; The geometric mean (95 percent confidence interval) concentration of GS-461203 in dried blood spots was compared between the pregnant cohort and 58 nonpregnant persons. The geometric mean (95 percent confidence interval) concentration of GS-461203 was 647 (571, 723) fmol/punch in the nonpregnant cohort; Test type: Other; Geometric mean ratio = .53, 95% CI 2-sided [.50 to .56] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

11. Secondary Outcome: Intracellular Concentration of GS-461203 From Dried Maternal Blood Spots at 6 Weeks
Description: Intracellular concentration of GS-461203, the active form of Sofosbuvir, from dried maternal blood spots measured 6 weeks after initiation of treatment
Time Frame: Approximately 6 weeks from initiation of treatment
Population: One participant discontinued study medication after the second daily dose
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/punch
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
fmol/punch | 340 [278 to 418]
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; [analysis description as in outcome 10, analysis 1]; Test type: Other; Geometric mean ratio = .53, 95% CI 2-sided [.49 to .58] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

12. Secondary Outcome: Intracellular Concentration of GS-461203 From Dried Maternal Blood Spots at 9 Weeks
Description: Intracellular concentration of GS-461203, the active form of Sofosbuvir, from dried maternal blood spots measured 9 weeks after initiation of treatment
Time Frame: Approximately 9 weeks from initiation of treatment
Population: One participant discontinued study medication after the second daily dose
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/punch
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 10
fmol/punch | 356 [275 to 461]
Statistical Analysis 1: Comparison: Sofosbuvir-Velpatasvir; [analysis description as in outcome 10, analysis 1]; Test type: Other; Geometric mean ratio = .55, 95% CI 2-sided [.48 to .64] — The pregnant cohort was the numerator, and the non-pregnant cohort was the denominator

13. Secondary Outcome: Quantity of Hepatitis C Virus in Maternal Plasma After Completion of Velpatasvir and Sofosbuvir Treatment
Description: Quantity of Hepatitis C RNA in maternal plasma measured at least 12 weeks after completion of Velpatasvir and Sofosbuvir treatment regimen
Time Frame: Approximately 24 weeks from initiation of treatment
Population: One participant discontinued study medication after the second daily dose, one participant was lost to follow-up.
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
copies/mL | NA [NA to NA] — Hepatitis C Viral RNA was not detectable in all participant samples; the lower limit of detection of the assay was 12 copies/mL.

14. Secondary Outcome: Number of Maternal and Infant Participants That Experience Adverse Events Related to Sofosbuvir/Velpatasvir
Description: Number of maternal and infant participants that experience an adverse event that is deemed related to Sofosbuvir/Velpatasvir by a study physician
Time Frame: Up to 16 weeks from initiation of treatment or 12 months from delivery
Population: There were 11 maternal-infant dyads
Measure: Count of Participants; unit: Participants
Groups:
- Sofosbuvir-Velpatasvir - Maternal Participants: One oral pill containing 400mg sofosbuvir and 100mg velpatasvir taken once daily for 12 weeks
- Sofosbuvir-Velpatasvir - Infant Participants: Infants born to mothers that took one oral pill containing 400mg sofosbuvir and 100mg velpatasvir taken once daily for 12 weeks during pregnancy
Arm/Group | Sofosbuvir-Velpatasvir - Maternal Participants | Sofosbuvir-Velpatasvir - Infant Participants
Number analyzed (Participants) | 11 | 11
Participants | 9 | 0

15. Secondary Outcome: Maternal Gestational Age at Delivery
Description: Maternal gestational age at delivery determined by medical record review
Time Frame: Up to 16 weeks from treatment initiation (at delivery)
Measure: Median (Full Range); unit: weeks
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 11
weeks | 39.00 [35.57 to 39.43]

16. Secondary Outcome: Infant Weight at Delivery
Description: Infant birth weight determined by medical record review
Time Frame: Up to 16 weeks from treatment initiation (at delivery)
Measure: Median (Full Range); unit: kg
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 11
kg | 2.90 [2.52 to 3.81]

17. Secondary Outcome: Frequency of Delivery Modes for Maternal Participants
Description: Frequency of delivery modes (spontaneous and assisted vaginal, scheduled and emergent cesarean section) for maternal participants determined by medical record review
Time Frame: Up to 16 weeks from treatment initiation (at delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 11
Participants
  Spontaneous vaginal delivery | 7
  Scheduled cesarean section | 3
  Emergent cesarean section | 1
  Assisted vaginal delivery | 0

18. Secondary Outcome: Number of Infant Participants With Congenital Anomalies
Description: Number of infant participants with congenital anomalies determined by medical record review for up to 12 months of age.
Time Frame: Up to 12 months from delivery
Population: Infant participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 11
Participants | 1

19. Secondary Outcome: Weight of Infant Participant at 1 to 3 Months
Description: Weight of infant participant measured at 1 to 3 months of age
Time Frame: Approximately 3 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Median (Full Range); unit: kg
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
kg | 5.6 [4.7 to 6.7]

20. Secondary Outcome: Weight of Infant Participant at 6 Months
Description: Weight of infant participant measured at 6 months of age
Time Frame: Approximately 6 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Median (Full Range); unit: kg
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
kg | 8.4 [6.7 to 9.8]

21. Secondary Outcome: Weight of Infant Participant at 12 Months
Description: Weight of infant participant measured at 12 months of age
Time Frame: Approximately 12 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Median (Full Range); unit: kg
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
kg | 10.6 [8.0 to 11.7]

22. Secondary Outcome: Length of Infant Participant at 1 to 3 Months
Description: Length of infant participant measured at 1 to 3 months of age
Time Frame: Approximately 3 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Median (Full Range); unit: cm
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
cm | 59.0 [53.0 to 65.0]

23. Secondary Outcome: Length of Infant Participant at 6 Months
Description: Length of infant participant measured at 6 months of age
Time Frame: Approximately 6 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Median (Full Range); unit: cm
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
cm | 67.0 [66.0 to 73.2]

24. Secondary Outcome: Length of Infant Participant at 12 Months
Description: Length of infant participant measured at 12 months of age
Time Frame: Approximately 12 months from delivery
Population: Two infant participants were lost to follow-up; length not assessed for 1 infant participant
Measure: Median (Full Range); unit: cm
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 8
cm | 76.2 [74.5 to 80.0]

25. Secondary Outcome: Head Circumference of Infant Participant at 1 to 3 Months
Description: Head circumference of infant participant measured at 1 to 3 months of age
Time Frame: Approximately 3 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Median (Full Range); unit: cm
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
cm | 39.5 [37.0 to 42.0]

26. Secondary Outcome: Head Circumference of Infant Participant at 6 Months
Description: Head circumference of infant participant measured at 6 months of age
Time Frame: Approximately 6 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Median (Full Range); unit: cm
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
cm | 43.4 [42.0 to 45.8]

27. Secondary Outcome: Head Circumference of Infant Participant at 12 Months
Description: Head circumference of infant participant measured at 12 months of age
Time Frame: Approximately 12 months from delivery
Population: Two infant participants were lost to follow-up; head circumference not assessed for 2 infant participants
Measure: Median (Full Range); unit: cm
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 7
cm | 46.4 [45.0 to 48.0]

28. Secondary Outcome: Quantity of Hepatitis C Virus in Infant Plasma at Birth
Description: Quantity of Hepatitis C viral RNA measured in infant plasma assessed at birth
Time Frame: Up to 16 weeks from treatment initiation (at delivery)
Population: One infant delivered at a non-study site hospital where Hepatitis C viral RNA in plasma was not assessed; 1 infant born maternal participant that did not complete study medication
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
copies/mL | NA [NA to NA] — Hepatitis C Viral RNA was not detectable in all participant samples; the lower limit of quantification for the assay was 12 copies/mL

29. Secondary Outcome: Quantity of Hepatitis C Virus in Infant Plasma at 1 to 3 Months
Description: Quantity of Hepatitis C viral RNA measured in infant plasma assessed at 1 to 3 months of age
Time Frame: Approximately 3 months from delivery
Population: Unable to obtain blood draw on 1 infant, 2 infants were lost to follow-up, 1 infant born maternal participant that did not complete study medication
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 7
copies/mL | NA [NA to NA] — Hepatitis C Viral RNA was not detectable in all participant samples; the lower limit of quantification for the assay was 15 copies/mL

30. Secondary Outcome: Quantity of Hepatitis C Virus in Infant Plasma at 6 Months
Description: Quantity of Hepatitis C viral RNA measured in infant plasma assessed at 6 months of age
Time Frame: Approximately 6 months from delivery
Population: Unable to obtain blood draw on 2 infants, 3 infants were lost to follow-up, 1 infant born maternal participant that did not complete study medication
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 5
copies/mL | NA [NA to NA] — Hepatitis C Viral RNA was not detectable in all participant samples; the lower limit of quantification for the assay was 15 copies/mL

31. Secondary Outcome: Quantity of Hepatitis C Virus in Infant Plasma at 12 Months
Description: Quantity of Hepatitis C viral RNA measured in infant plasma assessed at 12 months of age
Time Frame: Approximately 12 months from delivery
Population: Unable to obtain blood draw on 1 infant, 3 infants were lost to follow-up, 1 infant born maternal participant that did not complete study medication, Hepatitis C viral RNA assessment not required from 4 infants per protocol
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 2
copies/mL | NA [NA to NA] — Hepatitis C Viral RNA was not detectable in all participant samples; the lower limit of quantification for the assay was 12 copies/mL

32. Secondary Outcome: Number of Infant Participants Referred for Early Neurological Development Intervention
Description: Number of infant participants referred for early intervention based on neurological development assessments using Bayley Scales of Infant and Toddler Development. Infant participants with a Bayley's score of less than 6 on either cognitive, motor or language development assessments indicates an infant at risk for delayed development; Bayley's score ranges from 1 (extremely low) to 19 (very superior)
Time Frame: Approximately 12 months from delivery
Population: Two infant participants were lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 9
Participants | 1

33. Secondary Outcome: Percentage of Unbound Sofosbuvir Measured in Maternal Plasma
Description: Percentage of Sofosbuvir not bound to protein out of total protein- unbound and bound Sofosbuvir measured in maternal plasma samples. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation. At the 6-week visit, a single convenience blood sample was collected.
Time Frame: Approximately 9 weeks from initiation of maternal treatment
Population: Assay was not done.
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 0

34. Secondary Outcome: Percentage of Unbound Velpatasvir Measured in Maternal Plasma
Description: Percentage of Velpatasvir not bound to protein out of total protein- unbound and bound Velpatasvir measured in maternal plasma samples. Plasma samples were obtained pre-dose and at 0.5-, 1-, 2-, 3-, 4-, 5-, 8-, and 12- and 24 hours post-dose at the 3- and 9-week visits after treatment initiation. At the 6-week visit, a single convenience blood sample was collected.
Time Frame: Approximately 9 weeks from initiation of maternal treatment
Population: Assay was not done
Arm/Group | Sofosbuvir-Velpatasvir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months from initiation of treatment for maternal participants or 1 year from delivery for infants
Arm/Group | Sofosbuvir-Velpatasvir - Maternal Participants | Sofosbuvir-Velpatasvir - Infant Participants
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11 | 5/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sofosbuvir-Velpatasvir - Maternal Participants (N=11) | Sofosbuvir-Velpatasvir - Infant Participants (N=11)
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) — Renal calculi, obstructing with hydronephrosis
Clubfoot (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cryptorchidism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Transient tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Positive toxicology screen (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sofosbuvir-Velpatasvir - Maternal Participants (N=11) | Sofosbuvir-Velpatasvir - Infant Participants (N=11)
Headache (Nervous system disorders) | 4 (5) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hemorrhage, postpartum (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sciatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental abscess (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatitis, contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Fluid overload, postpartum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension, gestational (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Group B Streptococcus (Infections and infestations) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Opioid withdrawal (General disorders) | 1 (1) | 0 (0)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (11)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Jaundice (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vision screen, abnormal (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Croup (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dacrocystitis (Eye disorders) | 0 (0) | 1 (1)
Diaper dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eye nystagmus (Eye disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gross motor scores borderline to below average (Nervous system disorders) | 0 (0) | 1 (1)
Hand, foot and mouth disease (General disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nursemaid's elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasolacrimal duct obstruction (General disorders) | 0 (0) | 1 (1)
Oral thrush (Infections and infestations) | 0 (0) | 1 (1)
Orolabial Herpes Simplex Virus (Infections and infestations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory Syncytial Virus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Roseola (General disorders) | 0 (0) | 1 (1)
Seborrhea of scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sickle cell trait (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Temperature instability (General disorders) | 0 (0) | 1 (1)
Tibial torsion of lower legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urogenital candidiasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT04382404/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT04382404/ICF_002.pdf